CLINICAL TRIAL: NCT04402619
Title: Online Cognitive Behavior Therapy in Routine Addiction Care for Comorbid Sleep Problems in Alcohol Use Disorder
Brief Title: Online Cognitive Behavior Therapy for Comorbid Sleep Problems in Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Philip Lindner, Head of Research and Development, Maria Ungdom Clinic, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCS Sömnskola
Record Dates: First submitted 2020-04-14; First posted 2020-05-27 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Use Disorder; Insomnia; Sleep Disorder; Dyssomnias
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Dyssomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online CBT (Experimental): Ten modules with minimum therapist guidance
  Interventions: Behavioral: Cognitive behavior therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — The ten modules cover:
  * Psychoeducation about sleep, sleep problems, and associations with alcohol
  * How to keep and use a sleep diary
  * Sleep hygiene
  * Sleep compression
  * Cognitive restructuring
  * Emotional regulation
  * Preparing for the future
  Other Names: Sleep compression; Sleep hygiene

SUMMARY:
The main goal is to study the effects of internet-delivered cognitive behavioural therapy with minimum guidance for comorbid sleep problems in alcohol use disorder, in routine addiction care.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is highly prevalent and a major contributor to the global burden of disease. Insomnia symptoms are very common among individuals with AUD, including those in recovery, which may in turn promote alcohol relapse. Specialization and silo phenomena in healthcare organization, separating addiction from other types of psychiatric care, means that individuals with AUD and comorbid sleep problems often have difficulty accessing evidence-treatment for the latter. Offering online treatment for sleep problems to individuals enrolled in traditional routine addiction care is an attractive and pragmatic approach to offering parallel treatments covering the full clinical presentation, which has not yet been evaluated. This pilot and feasibility trial will recruit n=25 from patients in routine addiction care with comorbid sleep problems and AUD, who will complete an online, ten-module, CBT-based treatment program with minimum guidance for sleep problems, tailored for individuals with AUD.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patient at Stockholm Center for Dependency Disorders
* Diagnosed alcohol use disorder
* Self-rated sleep problem

Exclusion Criteria:

* Addiction to sedative or hypnotic medication
* Psychoactive medication not yet 3-month stable in dose
* Bipolar disorder
* Psychotic disorder
* Suicidality
* Periodic Limb Movement Disorder (PLMD)
* Sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Two-item Sleep Condition Indicator | Weeks 1 through 10 (max 15)
  Total score of the two-item SCI, assessing last-week symptoms. Administered on the treatment platform.

SECONDARY OUTCOMES:
Sleep Condition Indicator | Change from baseline (pre-treatment), post-treatment (primary endpoint, 10-15 weeks after baseline), and follow-up three months after baseline..
  Change in score on the full and regular SCI. Administered through the online survey tool connected to regular patient records system.
Daily sleep diary | Weeks 1 through 10 (max 15)
  Derived measures: last-week average sleep efficiency, time to fall asleep, time awake at night, total sleep time.
Daily alcohol diary | Weeks 1 through 10 (max 15)
  Total consumed standard units of alcohol per week, during day and before bedtime
Alcohol Use Disorders Identification Test (AUDIT) | Change from baseline (pre-treatment), post-treatment (primary endpoint, 10-15 weeks after baseline), and follow-up three months after baseline..
  Total score
Drug Use Disorders Identification Test (DUDIT) | Change from baseline (pre-treatment), post-treatment (primary endpoint, 10-15 weeks after baseline), and follow-up three months after baseline..
  Total score
Patient Health Questionnaire-9 (PHQ9) | Change from baseline (pre-treatment), post-treatment (primary endpoint, 10-15 weeks after baseline), and follow-up three months after baseline..
  Total score
Health-related quality of life (EQ5D) | Change from baseline (pre-treatment), post-treatment (primary endpoint, 10-15 weeks after baseline), and follow-up three months after baseline..
  Total score

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lindner, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Stockholm Addiction eClinic (eStöd, Beroendecentrum Stockholm), Stockholm
  - Stockholm Centre for Dependency Disorders, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Raw outcomes, with any other identifiable information, may be shared under the conditions described below.
Time Frame: Requests for data will be accepted upon publication of trial, and for ten years after.
Access Criteria: Signed data sharing agreement.

REFERENCES:
- [Background] Kaldo V, Jernelov S, Blom K, Ljotsson B, Brodin M, Jorgensen M, Kraepelien M, Ruck C, Lindefors N. Guided internet cognitive behavioral therapy for insomnia compared to a control treatment - A randomized trial. Behav Res Ther. 2015 Aug;71:90-100. doi: 10.1016/j.brat.2015.06.001. Epub 2015 Jun 3. PMID 26091917